CLINICAL TRIAL: NCT07317206
Title: Effects of Single Dose of Ayahuasca or Esketamine on Posttraumatic Stress Disorder: a Randomized, Double-blinded Study
Brief Title: Ayahuasca, Esketamine and PTSD
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Rafael Guimarães dos Santos, PhD, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 55068322.2.0000.5440
Record Dates: First submitted 2025-12-19; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Posttraumatic Stress Disorder (PTSD)
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Esketamine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ayahuasca (Experimental): oral ayahuasca
  Interventions: Drug: Ayahuasca
- esketamine (Active Comparator): oral esketamine
  Interventions: Drug: Esketamine

INTERVENTIONS:
Drug: Ayahuasca — oral ayahuasca
  Arms: Ayahuasca
Drug: Esketamine — oral esketamine
  Arms: esketamine

SUMMARY:
Double-blind, randomized trial comparing a single dose of oral ayahuasca or esketamine in patients with posttraumatic stress disorder.

ELIGIBILITY:
Inclusion Criteria:

* posttraumatic stress disorder

Exclusion Criteria:

* psychiatric and other medical comorbidities

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-12-20 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Posttraumatic Stress Disorder Checklist for DSM-5 | From enrollment to the end of treatment at 3 weeks
  higher scores mean a worse outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital das Clínicas da FMRP-USP, Ribeirão Preto, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No